CLINICAL TRIAL: NCT00141869
Title: MEG Study of Altered Sensory Processing in Tourette Syndrome: An Exploration of Sensory Tics
Brief Title: Brain Activity Associated With Tics in Patients With Tourette Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050230; 05-N-0230
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-09-06

CONDITIONS: Tourette Syndrome
Keywords: Sensory Processing; Magnetoencephalogram; Tourete Syndrome; Trigeminal Nerve; Tics; TS; Healthy Volunteer; HV
MeSH Terms: conditions — Tourette Syndrome; Tics

SUMMARY:
This study will examine brain activity associated with the involuntary urges or uncontrolled movements, called "tics," experienced by people who have Tourette syndrome (TS). Before people with TS actually develop a tic, whether it is a movement or a vocal tic (like a cough or bark), they feel the urge to tic. This study will look at brain activity during the time of this urge and how brain activity may differ in people with TS and without TS.

Healthy normal volunteers and patients with TS between 14 and 65 years of age may be eligible for this study. Patients must have sensory tics in the facial region and must experience at least a moderate premonitory urge. Candidates are screened with a medical history, brief physical examination, and a questionnaire.

Participants undergo the following procedures:

* Magnetoencephalography (MEG): This test records magnetic field changes produced by brain activity. During the test, the subjects are seated in the MEG recording room and a cone containing magnetic field detectors is lowered onto their head. Electrodes (small metal disks) are placed on both sides of the face near the jaw. The recording may be made while the subject receives small currents from the electrodes on the jaw. Subjects may be asked a few questions about what they felt during the procedure.
* Magnetic resonance imaging (MRI): This test uses a strong magnetic field and radio waves to obtain images of body organs and tissues. During the procedure, the subject lies on a table that can slide in and out of the scanner-a metal cylinder. Subjects may be asked to lie still for up to 30 minutes at a time. They can communicate with the staff at any time during the scan.
* Somatosensory evoked responses: This test examines how sensory information travels form the nerves to the spinal cord and brain in the nervous system. An electrode placed on the arm, leg, or face delivers a small electrical stimulus that may tingle and cause a twitch of a hand, foot, or face muscle. Additional electrodes may sometimes be placed on the scalp, neck, and over the collarbone to record how the impulse from the stimulus travels over nerve pathways.

Patients in the study are contacted for follow-up after the study. Follow-up will be conducted by phone or email, according to the patients' convenience, and will consist of reaffirming that there were no adverse events.

DETAILED DESCRIPTION:
OBJECTIVES:

This study will examine the spatiotemporal dynamics of sensory tics in patients with Tourette syndrome (TS). We will also investigate the possible existence of a sensory gating problem. By investigating somatosensory evoked responses from stimulation of the trigeminal nerve (tSERs) on affected versus unaffected sides of the face, we hope to identify differences in the SER waveforms that suggest sensory abnormalities. We will use a series of short trains of stimulations on the affected side to examine habituation, subsequently performing a time-

frequency analysis to seek indicators of decreased sensory gating. This study will examine, specifically:

Whether the cortical neurocircuitry involved in the elicitation of tSERs differs in patients with tic disorders from controls.

If SERs differ in a sensory tic facial region of patients, compared to the same spot on an unaffected side of the face.

Whether in controls and patients with sensory tics on both sides of their body, tSERs on both sides of the face are symmetrical.

If there is a lack of habituation in tic patients to tSERs in a short-train click paradigm, compared to controls.

The location for sources of abnormalities in either paradigm.

STUDY POPULATION:

Twenty patients and 10 control subjects will be studied. Subjects can be of any race, gender, handedness, or age between 14 and 65 years.

DESIGN:

This study will compare tSERs in normal volunteers to those in TS patients. Patients with bilateral sensory tics will be contrasted with those who have unilateral sensory tics, comparing power of the response at latencies on affected versus unaffected sides. Subjects will be seated in the MEG and instructed to "feel the delivered sensation, and try not to tic for seventy seconds, without counting". The trigeminal nerve will be electrically stimulated at 0.25 Hz for 30 seconds, which will be followed by head localization and subsequent rest for tic release. To evaluate sensory gating, the design is similar except the trigeminal stimulation will occur in short trains. Patients will be surveyed to determine if the instructions intensified sensory tics.

OUTCOME MEASURES:

We will compare the power of averaged tSERs at latencies, comparing face sides in patients and comparing patients' active face side with controls' dominant face side. The power of frequency components at latencies will be considered. We will locate the sources of differential tSER activity.

ELIGIBILITY:
* INCLUSION CRITERIA FOR NORMAL VOLUNTEERS:

Subjects will be normal volunteers with no history of neurological disorders; they will be screened in the NINDS Movement Disorders Outpatient Clinic, and will have a neurological and physical examination.

Subjects will be male or female, in age ranges 14 to 65 years old.

INCLUSION CRITERIA FOR PATIENTS:

Patients ages 14 to 65 with a clinical diagnosis of tourette syndrome or chronic motor tic disorder as defined by DSM-IV-TR and evaluation of tic severity using the Yale Tic Scale (YGTSS). This criterion will be established by preliminary screening in the NINDS Movement Disorders Outpatient Clinic. Structure Clinical Interview for (DSMIV SCID) will be administered to all subjects to ensure that strict DSM-IV criteria for Tourette syndrome have been met and to assess for possible comorbid psychiatric disorders.

Patients with at least moderate premonitory urge, as evaluated with the PUTS.

Patients with sensory tics, either bilaterally or unilaterally, in the facial region.

EXCLUSION CRITERIA FOR PATIENTS AND NORMAL VOLUNTEERS:

Cardiac pacemaker / cardiac or neural defibrillators.

Metal fragments in the eyes.

Metal plates, pins, or bolts in the head.

Any magnetic implantation / implantations made from iron (ferrous products).

Hearing problems.

Problems using response devices.

Subjects younger than 14 or older than 65 years.

Subjects with 1 ) major depression, 2) bipolar disorder, or 3) psychotic disorder.

Subjects taking benzodiazepines, anti-depressant or neuroleptic medications.

Subjects with major acute or chronic illness, or subjects for whom sitting in a still position for an extended period of time would trigger or exacerbate a preexisting condition or cause any undue harm or discomfort.

Pregnant women (steroidal hormones have been shown to influence EEG (Rupprecht et al., 2001).

Patients with severe head tics or subjects who are unable to hold their head still in a scanner for at least 70 seconds.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-08-30; Study Completion 2007-09-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bliss J. Sensory experiences of Gilles de la Tourette syndrome. Arch Gen Psychiatry. 1980 Dec;37(12):1343-7. doi: 10.1001/archpsyc.1980.01780250029002. PMID 6934713